CLINICAL TRIAL: NCT00115115
Title: Prospective Randomized Trial to Evaluate the Efficacy of Donor Preconditioning With Dopamine on Initial Graft Function After Kidney Transplantation
Brief Title: Donor Dopamine and Initial Graft Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitätsmedizin Mannheim (Other)
Collaborators: Eurotransplant International Foundation, Leiden, The Netherlands (Other); Regional Organ Procurement Organization (DSO), Baden-Wuerttemberg, Germany (Other); Regional Organ Procurement Organization (DSO), Bavaria, Germany (Other); Novartis (Industry)
Responsible Party: Peter Schnuelle, MD, University Hospital Mannheim, Dept. of Medicine V, Theodor Kutzer Ufer 1-3, 68135 Mannheim, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3074_KAC03.wpd
Record Dates: First submitted 2005-06-20; First posted 2005-06-21 (Estimated); Last update posted 2009-04-23 (Estimated); Status verified 2009-04

CONDITIONS: Kidney Transplantation; ESRD
Keywords: Donor dopamine; Immediate graft function; Kidney transplantation
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Dopamine infusion to brain dead organ donors — Dopamine infusion administered at a dosage of 4µg/kg/min starting after brain death has been proven until to surgical procurement of the kidneys

SUMMARY:
Donor pre-treatment with dopamine reduces injury to the kidney graft with consequences on the clinical performance immediately after transplantation: Donor dopamine reduces the requirement of dialysis post transplant, and results in renal function improvements.

The purpose of the study is to investigate the potentially therapeutic impact of donor preconditioning with low dose dopamine in human renal transplant recipients from a brain dead donor.

DETAILED DESCRIPTION:
During the transplantation process, the kidney graft is exposed to numerous events which may in turn lead to function deteriorations. In particular, factors related with brain death, like hemodynamic instability and systemic release of cytokines, cold preservation upon harvesting, and reperfusion injury accumulate in harm conveying a pro-inflammatory state to the graft before transplantation. Early graft dysfunction has long-term consequences. Renal transplants with delayed graft function and acute rejection have a greater incidence of chronic dysfunction. Allorecognition is induced when the host immune system detects alloantigens in the context of danger signals. Reducing danger signals through medical donor management may therefore have a considerable impact on the transplantation outcomes.

In a case control study from the Transplantation Center of Mannheim, Germany, donor use of both dopamine and noradrenaline during intensive care before organ retrieval was associated with less acute rejection episodes after transplantation and resulted in superior long-term graft survival. Donor employment of catecholamines remained predictive of an improved graft survival probability even after controlling for various confounding factors like age, gender, cold ischemia, HLA matching and immunosuppressive medication. This observation has been confirmed by a larger retrospective cohort study based on the Eurotransplant registry, including 2404 kidney transplants performed at 47 renal transplantation centers in 1993. The salutary effect on the graft function rate at 4 years exhibited a dose-response relationship and compared in quantitative terms with prospective HLA matching on class I or II antigens. Besides these long-term benefits, donor preconditioning with dopamine is associated with improvements of immediate graft function after kidney transplantation. Donor dopamine was associated with less requirement of hemodialysis and more rapid recovery of graft function posttransplant in a single centre study involving 254 consecutive renal transplant recipients.

Implementing dopamine as a therapeutic tool in the management of cadaver kidney donors may have a major impact on both immediate graft function and long-term graft survival without adverse side effects for the recipients.

ELIGIBILITY:
Inclusion Criteria:

Donors:

* Brain death confirmed
* Given consent to organ donation
* Current s-creatinine < 2mg/dl
* On admission s-creatinine < 1.3mg/dl

Recipients:

* Age over 18 years
* Placed on the waiting list
* Organ allocation according to ET standards

Exclusion Criteria:

Donors:

* Application of dopamine/dobutamine/adrenaline
* Application of noradrenaline > 0.4µg/kg*min
* Hemodynamic instability

Recipients:

* Refusal to participate in study /data analysis
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 487 (Actual)
Dates: Start 2004-03; Primary Completion 2007-12 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Requirement of hemodialysis post-transplant | within 1 week after surgery

SECONDARY OUTCOMES:
Incidence and severity of acute rejection episodes | within the first 30 days (plus minus 3 days) after surgery
S-creatinine on days 1-7 post transplant | within the first week after transplantation
Patient and graft survival | after 12, 24 and 36 months post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schnuelle, MD, Principal Investigator — Universitätsmedizin Mannheim; Fokko J van der Woude, MD, PhD, Study Chair — Universitätsmedizin Mannheim; Werner Lauchart, MD, Study Director — Organ procurement organization (DSO) of Baden-Wuerttemberg; Detlef Boesebeck, MD, Study Director — Organ procurement organization (DSO) of Bavaria
Locations (1):
- University Hospital Mannheim, Mannheim, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Schnuelle P, Yard BA, Braun C, Dominguez-Fernandez E, Schaub M, Birck R, Sturm J, Post S, van der Woude FJ. Impact of donor dopamine on immediate graft function after kidney transplantation. Am J Transplant. 2004 Mar;4(3):419-26. doi: 10.1111/j.1600-6143.2004.00331.x. PMID 14961996
- [Background] Yard B, Beck G, Schnuelle P, Braun C, Schaub M, Bechtler M, Gottmann U, Xiao Y, Breedijk A, Wandschneider S, Losel R, Sponer G, Wehling M, van der Woude FJ. Prevention of cold-preservation injury of cultured endothelial cells by catecholamines and related compounds. Am J Transplant. 2004 Jan;4(1):22-30. doi: 10.1046/j.1600-6143.2003.00268.x. PMID 14678031
- [Background] Schnuelle P, Berger S, de Boer J, Persijn G, van der Woude FJ. Effects of catecholamine application to brain-dead donors on graft survival in solid organ transplantation. Transplantation. 2001 Aug 15;72(3):455-63. doi: 10.1097/00007890-200108150-00017. PMID 11502976
- [Background] Schnuelle P, Lorenz D, Mueller A, Trede M, Van Der Woude FJ. Donor catecholamine use reduces acute allograft rejection and improves graft survival after cadaveric renal transplantation. Kidney Int. 1999 Aug;56(2):738-46. doi: 10.1046/j.1523-1755.1999.00567.x. PMID 10432416
- [Derived] Benck U, Jung M, Kruger B, Grimm A, Weiss C, Yard BA, Lehner F, Kiessling A, Fischer L, Gallinat A, Kleespies A, Lorf T, Sucher R, Monch C, Scherer MN, Rahmel A, Schemmer P, Kramer BK, Schnuelle P. Donor Dopamine Does Not Affect Liver Graft Survival: Evidence of Safety From a Randomized Controlled Trial. Liver Transpl. 2018 Oct;24(10):1336-1345. doi: 10.1002/lt.25301. PMID 30102825
- [Derived] Schnuelle P, Benck U, Kramer BK, Yard BA, Zuckermann A, Wagner F, Szabo G, Borggrefe M, Karck M, Gummert J. Impact of Donor Core Body Temperature on Graft Survival After Heart Transplantation. Transplantation. 2018 Nov;102(11):1891-1900. doi: 10.1097/TP.0000000000002337. PMID 29994980
- [Derived] Schnuelle P, Mundt HM, Druschler F, Schmitt WH, Yard BA, Kramer BK, Benck U. Impact of spontaneous donor hypothermia on graft outcomes after kidney transplantation. Am J Transplant. 2018 Mar;18(3):704-714. doi: 10.1111/ajt.14541. Epub 2017 Nov 22. PMID 29027352
- [Derived] Schnuelle P, Schmitt WH, Weiss C, Habicht A, Renders L, Zeier M, Druschler F, Heller K, Pisarski P, Banas B, Kramer BK, Jung M, Lopau K, Olbricht CJ, Weihprecht H, Schenker P, De Fijter JW, Yard BA, Benck U. Effects of Dopamine Donor Pretreatment on Graft Survival after Kidney Transplantation: A Randomized Trial. Clin J Am Soc Nephrol. 2017 Mar 7;12(3):493-501. doi: 10.2215/CJN.07600716. Epub 2017 Feb 17. PMID 28213388
- [Derived] Benck U, Gottmann U, Hoeger S, Lammert A, Rose D, Boesebeck D, Lauchart W, Birck R, Weiss C, Kramer BK, Yard BA, Schnuelle P. Donor desmopressin is associated with superior graft survival after kidney transplantation. Transplantation. 2011 Dec 15;92(11):1252-8. doi: 10.1097/TP.0b013e318236cd4c. PMID 22067309
- [Derived] Benck U, Hoeger S, Brinkkoetter PT, Gottmann U, Doenmez D, Boesebeck D, Lauchart W, Gummert J, Karck M, Lehmkuhl HB, Bittner HB, Zuckermann A, Wagner F, Schulz U, Koch A, Bigdeli AK, Bara C, Hirt S, Berchtold-Herz M, Brose S, Herold U, Boehm J, Welp H, Strecker T, Doesch A, Birck R, Kramer BK, Yard BA, Schnuelle P. Effects of donor pre-treatment with dopamine on survival after heart transplantation: a cohort study of heart transplant recipients nested in a randomized controlled multicenter trial. J Am Coll Cardiol. 2011 Oct 18;58(17):1768-77. doi: 10.1016/j.jacc.2011.05.060. PMID 21996389
- [Derived] Schnuelle P, Gottmann U, Hoeger S, Boesebeck D, Lauchart W, Weiss C, Fischereder M, Jauch KW, Heemann U, Zeier M, Hugo C, Pisarski P, Kramer BK, Lopau K, Rahmel A, Benck U, Birck R, Yard BA. Effects of donor pretreatment with dopamine on graft function after kidney transplantation: a randomized controlled trial. JAMA. 2009 Sep 9;302(10):1067-75. doi: 10.1001/jama.2009.1310. PMID 19738091